CLINICAL TRIAL: NCT07192172
Title: Enhanced Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma Post-Trans-arterial Chemoembolization: A Prospective Study Using Twin Internally Cooled-Perfusion Electrodes
Brief Title: Enhanced Radiofrequency Ablation for Recurrent HCC Post-TACE Using Twin Internally Cooled-Perfusion Electrodes
Acronym: ERFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH 1611124811; No. 06-2017-0260 (Other Grant/Funding Number: RF Medical)
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Recurrent HCC; Ablation Techniques, RFA
Keywords: Recurrent Hepatocellular carcinoma; Radiofrequency ablation; Bipolar; HCC; Image guidance; Local tumor progression
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Single Group Assignment, radiofrequency ablation (NT-RFA) using twin cooled wet (TCW) electrodes in patients experiencing recurrent hepatocellular carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Bipolar RFA using TICP electrodes (Other): All participants receive bipolar RFA treatment using TICP electrodesTreatment is conducted under real-time ultrasound-CT/MR fusion guidance
  Interventions: Device: Bipolar radiofrequency ablation using twin internally cooled perfusion electrodes

INTERVENTIONS:
Device: Bipolar radiofrequency ablation using twin internally cooled perfusion electrodes — Device: Twin Internally Cooled-Perfusion (TICP) Electrodes
  Two 17-gauge internally cooled-perfusion electrodes Multichannel RF generator (RF Medical Co., Seoul, Korea) Bipolar mode application Saline perfusion rate: approximately 1 cc/min

SUMMARY:
This single-center, prospective study evaluates the therapeutic outcomes of saline-augmented bipolar radiofrequency ablation (RFA) with twin internally cooled-perfusion (TICP) electrodes for treating recurrent hepatocellular carcinoma (HCC) following trans-arterial chemoembolization (TACE).

DETAILED DESCRIPTION:
The primary endpoint was defined as the 2-year cumulative incidence of LTP of the ablation index tumor, measured from the RFA date to first LTP occurrence. Secondary endpoints encompassed technical success rate, technique efficacy, RFA procedure characteristics, and progression-free survival (PFS) post-RFA. Data collection continued through July 31, 2020.

Between September 2017 and January 2019, we screened patients with recurrent HCC after TACE for study eligibility (Figure 1). Inclusion criteria specified: a) age between 20 and 85 years, b) Child-Pugh Class A liver function, and c) radiologically confirmed locally recurrent HCC following conventional TACE treatment.

Recurrent HCC was defined as the appearance of arterially enhancing tumor at the edge of the treated tumor, after at least one contrast-enhanced follow-up study had documented adequate lipiodol uptake and absence of viable tissue in the target tumor and surrounding ablation margin, as assessed using modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria (5). Recurrence was primarily diagnosed using contrast-enhanced multiphasic CT (n=73) or MRI (n=27). The exclusion criteria consisted of the following: a) more than three HCC nodules, b) tumors with an abutment length of ≥5 mm to the main hepatic veins or the first branches of the main portal vein, c) HCC nodules measuring 3 cm or larger, d) platelet count ≤50,000/mm³ or international normalized ratio prolongation ≥50%, e) extrahepatic metastasis or vascular invasion, f) Child-Pugh class B or C, g) poor performance status of Eastern Cooperative Oncology Group-performance status scale 3 or higher, and h) cases with poor acoustic window or inability to achieve percutaneous access.

RFA procedures RFA procedures were conducted under real-time US/CT/MR fusion guidance (Samsung, Navigator-GE & Siemens, PercuNav-Phillips) with conscious sedation by a radiologist (J.M.L.) with 26 years of clinical experience in RFA. The procedure utilized two 17-gauge internally cooled-perfusion electrodes and a multichannel RF generator (RF Medical Co., Seoul, Korea) in bipolar mode. In the bipolar mode, the current flows between the pair of electrodes and through this, a higher current density is maintained (12). The TICP electrodes featured two side holes (0.02 mm in diameter) on the active tips, through which 0.9% isotonic saline was perfused at approximately 1 cc/min for tissue perfusion and electrode cooling (Figure 2). A peristaltic pump (VIVA Pump; STARmed) maintained the active tip temperature at 20-25°C by circulating chilled normal saline. The ablation protocol aimed to completely ablate the entire tumor, including both the post-TACE area and locally recurrent lesion, while achieving a 5-10 mm wide ablation margin (13). Technical parameters, including current, impedance, power output, and total delivered energy, were continuously monitored. For subcapsular tumors, artificial ascites using 5% dextrose solution was employed in 80 patients (80.0%) to prevent organ damage and was subsequently aspirated post-procedure (14).

Evaluation of Procedure and Follow-up Technical success was defined as complete tumor treatment with full coverage by ablative margin ≥5 mm on immediate follow-up CT (15). One month after RFA, participants underwent contrast-enhanced CT (n=92) or MRI (n=8), serum alpha-fetoprotein measurements, and liver function tests. At this time point, technique efficacy was assessed, defined as complete ablation of macroscopic tumor (15). Ablation volume was quantified using the one-month follow-up images by measuring three orthogonal diameters (x, y, z) and calculating the volume using the formula: V=4/3 π× x × y × z (16). Follow-up imaging included contrast-enhanced multiphasic CT or MRI at 3, 6, and 12 months in the first year, followed by imaging every 3 months thereafter until study completion on July 31, 2020. LTP was defined as the appearance of enhancement at the ablation margin on contrast-enhanced imaging (11, 17). PFS encompassed all forms of disease progression, including not only LTP but also intrahepatic remote recurrence (defined as the presence of HCC in the liver at a site not contiguous with the ablation zone) and extrahepatic metastasis (defined as the spread of HCC to locations outside the liver) (11).

Statistical Analysis Statistical analysis was performed using SPSS (version 27) and MedCalc (version 20.0.23). Continuous variables were analyzed using Mann-Whitney U tests, and categorical variables using chi-square or Fisher's exact tests. Technical success, technique efficacy, and LTP rates were analyzed using per-patient data. Kaplan-Meier methods were employed for time-to-event analysis, with statistical significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-85 years Child-Pugh Class A liver function Radiologically confirmed locally recurrent HCC following conventional TACE treatment Recurrent HCC defined as arterially enhancing tumor at the edge of treated tumor

Exclusion Criteria:

* More than three HCC nodules Tumors with ≥5 mm abutment length to main hepatic veins or first branches of main portal vein HCC nodules ≥3 cm Platelet count ≤50,000/mm³ or INR prolongation ≥50% Extrahepatic metastasis or vascular invasion Child-Pugh class B or C ECOG performance status ≥3 Poor acoustic window or inability to achieve percutaneous access

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
2-year cumulative incidence of local tumor progression (LTP) | Time Frame: 2 years
  2-year cumulative incidence of local tumor progression (LTP) Description: LTP defined as the appearance of enhancement at the ablation margin on contrast-enhanced imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hosptial, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Timing:, after publication Access Process: submission of a request to the authors). Conditions for Use: for academic purposes only
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: Conditions for Use: for academic purposes only
URL: http://cris.snuh.org

REFERENCES:
- [Background] Choi JW, Lee JM, Lee DH, Yoon JH, Kim YJ, Lee JH, Yu SJ, Cho EJ. Radiofrequency Ablation Using a Separable Clustered Electrode for the Treatment of Hepatocellular Carcinomas: A Randomized Controlled Trial of a Dual-Switching Monopolar Mode Versus a Single-Switching Monopolar Mode. Korean J Radiol. 2021 Feb;22(2):179-188. doi: 10.3348/kjr.2020.0134. Epub 2020 Jul 22. PMID 32729269
- Available data/document: Study Protocol: No. 1611-124-811 — http://cris.snuh.org — http://cris.snuh.org